CLINICAL TRIAL: NCT02466516
Title: A Phase 2, Randomized, Open Label Study Evaluating the Safety, Tolerability, and Efficacy of GS-4997 Alone or in Combination With Simtuzumab (SIM) in Subjects With Nonalcoholic Steatohepatitis (NASH) and Fibrosis Stages F2-F3
Brief Title: Safety, Tolerability, and Efficacy of GS-4997 Alone or in Combination With Simtuzumab (SIM) in Adults With Nonalcoholic Steatohepatitis (NASH) and Fibrosis Stages F2-F3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-384-1497
Record Dates: First submitted 2015-06-05; First posted 2015-06-09 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-05

CONDITIONS: Non-Alcoholic Steatohepatitis (NASH)
Keywords: GS-4997; Non-alcoholic fatty liver disease (NAFLD); Fibrosis; Simtuzumab (SIM); Apoptosis signal-regulating kinase 1; ASK1 inhibitor
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fibrosis | interventions — simtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- SEL 6 mg (Experimental): Selonsertib (SEL) 6 mg for 24 weeks.
  Interventions: Drug: SEL
- SEL 18 mg (Experimental): SEL 18 mg for 24 weeks.
  Interventions: Drug: SEL
- SEL 6 mg+SIM 125 mg (Experimental): SEL 6 mg plus SIM 125 mg for 24 weeks.
  Interventions: Drug: SEL; Biological: SIM
- SEL 18 mg+SIM 125 mg (Experimental): SEL 18 mg plus SIM 125 mg for 24 weeks.
  Interventions: Drug: SEL; Biological: SIM
- SIM 125 mg (Experimental): SIM 125 mg for 24 weeks.
  Interventions: Biological: SIM

INTERVENTIONS:
Drug: SEL — SEL tablet administered orally once daily
  Other Names: GS-4997
  Arms: SEL 18 mg; SEL 18 mg+SIM 125 mg; SEL 6 mg; SEL 6 mg+SIM 125 mg
Biological: SIM — Simtuzumab (SIM) 125 mg/mL single-dose vials administered subcutaneously once weekly
  Other Names: GS-6624
  Arms: SEL 18 mg+SIM 125 mg; SEL 6 mg+SIM 125 mg; SIM 125 mg

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of GS-4997 (selonsertib [SEL]) alone or in combination with simtuzumab (SIM) in adults with nonalcoholic steatohepatitis (NASH) and fibrosis stages F2-F3. Participants will be randomized in a 2:2:1:1:1 ratio to 1 of 5 study treatment arms.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and non-pregnant, non-lactating females
* Evidence of NASH with fibrosis on biopsy

Key Exclusion Criteria:

* Cirrhosis of the liver (e.g. Brunt/Kleiner score of F4)
* Other causes of liver disease including viral hepatitis and alcoholic liver disease
* Any history of decompensated liver disease, including ascites, hepatic encephalopathy or variceal bleeding
* History of liver transplantation
* Alcohol consumption greater than 21 oz/week for males or 14 oz/week for females (1 oz/30 mL of alcohol is present in 1 12 oz/360 mL beer, 1 4 oz/120 mL glass of wine, and a 1 oz/30 mL measure of 40% proof alcohol)

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-06-08 (Actual); Primary Completion 2016-10-11 (Actual); Study Completion 2016-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (28):
- United States (26):
  - Stanford University Medical Center, Palo Alto, California
  - University of California San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado Denver, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Mercy Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Kansas City Research Institute, Kansas City, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburg Medical Center, Pittsburgh, Pennsylvania
  - Texas Clinical Research Institute, Arlington, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - CHI St. Luke's Health Baylor College of Medicine, Houston, Texas
  - Brooke Army Medical Center Ft. Sam, Houston, Texas
  - Digestive Research Center, Live Oak, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Mary Immaculate Hospital, Newport News, Virginia
  - St. Mary's Hospital, Richmond, Virginia
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Toronto Liver Centre, Toronto, Ontario

REFERENCES:
- [Result] Loomba R, Lawitz E, Mantry PS, Jayakumar S, Caldwell SH, Arnold H, et al. GS-4997, an inhibitor of apoptosis signal-regulating kinase (ASK1), alone or in combination with simtuzumab for the treatment of nonalcoholic steatohepatitis (NASH): a randomized, phase 2 trial. Hepatol 2016; 64 (6S): 1119A-1120A.
- [Result] Diehl AM, French D, Xu R, et al. Treatment with selonsertib, an inhibitor of apoptosis signal-regulating kinase 1, hepatic phospho-p38 expression and markers of hepatocellular apoptosis and necrosis in patients with nonalcoholic steatohepatitis. J Hepatol 2017;66:S51. PS-090.
- [Result] Middleton MS, Lawitz E, Jayakumar S, et al. Hepatic proton density fat fraction correlates with histologic measures of steatosis and is responsive to change in those measures in a multi-center nonalcoholic steatohepatitis clinical trial. J Hepatol 2017;66:S668. SAT-483.
- [Result] Loomba R, Lawitz E, Ghalib R, et al. Longitudinal changes in liver stiffness by magnetic resonance elastography (MRE), liver fibrosis, and serum markers of fibrosis in a multi-center clinical trial in nonalcoholic steatohepatitis (NASH). J Hepatol 2017;66:S671. SAT-489.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States and Canada. The first participant was screened on 08 June 2015.The last study visit occurred on 11 October 2016.
Pre-assignment Details: 242 participants were screened.
Groups:
- SEL 6 mg: Selonsertib (SEL) 6 mg tablet once daily for 24 weeks.
- SEL 18 mg: SEL 18 mg tablet once daily for 24 weeks.
- SEL 6 mg+SIM 125 mg: SEL 6 mg tablet once daily plus simtuzumab (SIM) 125 mg/mL administered subcutaneously once weekly for 24 weeks.
- SEL 18 mg+SIM 125 mg: SEL 18 mg tablet once daily plus SIM 125 mg/mL administered subcutaneously once weekly for 24 weeks.
- SIM 125 mg: SIM 125 mg/mL administered subcutaneously once weekly for 24 weeks.
Period: Overall Study
Arm/Group | SEL 6 mg | SEL 18 mg | SEL 6 mg+SIM 125 mg | SEL 18 mg+SIM 125 mg | SIM 125 mg
Started | 20 | 22 | 10 | 10 | 10
Completed | 16 | 21 | 9 | 10 | 10
Not Completed | 4 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Withdrew Consent | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | SEL 6 mg | SEL 18 mg | SEL 6 mg+SIM 125 mg | SEL 18 mg+SIM 125 mg | SIM 125 mg | Total
Number analyzed (Participants) | 20 | 22 | 10 | 10 | 10 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11.5) | 56 (9.0) | 52 (9.7) | 51 (11.1) | 57 (7.7) | 54 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 9 | 7 | 6 | 50
  Male | 7 | 7 | 1 | 3 | 4 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 5 | 2 | 1 | 22
  Not Hispanic or Latino | 13 | 15 | 5 | 8 | 9 | 50
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 3 | 1 | 0 | 1 | 0 | 5
  Race: Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  Race: White | 17 | 19 | 10 | 9 | 10 | 65
  Race: Not Permitted | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 1 | 0 | 1 | 1 | 6
  United States | 17 | 21 | 10 | 9 | 9 | 66

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Treatment-Emergent Adverse Events (TEAEs), Treatment-Emergent Serious Adverse Events (SAEs), and Any Grade ≥ 1 Laboratory Abnormality
Description: Treatment-emergent events began on or after the first dosing date up to 30 days after the last dosing date or led to premature discontinuation of study drug. The severity of laboratory abnormalities was assessed as Grade 0, 1 (mild), 2 (moderate), 3 (severe), or 4 (potentially life threatening) using the Common Terminology Criteria for Adverse Events (CTCAE), version 4.03.
Time Frame: Baseline up to last dose plus 30 days (up to Week 28)
Population: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | SEL 6 mg | SEL 18 mg | SEL 6 mg+SIM 125 mg | SEL 18 mg+SIM 125 mg | SIM 125 mg
Number analyzed (Participants) | 20 | 22 | 10 | 10 | 10
Participants
  TEAEs | 17 | 15 | 9 | 9 | 7
  SAEs | 2 | 2 | 0 | 1 | 0
  Any Grade ≥ 1 Laboratory Abnormality | 17 | 21 | 9 | 10 | 8

2. Primary Outcome: Number of Participants Who Prematurely Discontinued Study Drug or Study Due to Adverse Events
Time Frame: Baseline up to follow up visit (Week 28)
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | SEL 6 mg | SEL 18 mg | SEL 6 mg+SIM 125 mg | SEL 18 mg+SIM 125 mg | SIM 125 mg
Number analyzed (Participants) | 20 | 22 | 10 | 10 | 10
Participants
  Discontinued Study Drug | 1 | 2 | 0 | 0 | 0
  Discontinued Study | 1 | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to last dose plus 30 days (up to Week 28)
Description: Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | SEL 6 mg | SEL 18 mg | SEL 6 mg+SIM 125 mg | SEL 18 mg+SIM 125 mg | SIM 125 mg
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 2/20 | 2/22 | 0/10 | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 17/20 | 14/22 | 9/10 | 9/10 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SEL 6 mg (N=20) | SEL 18 mg (N=22) | SEL 6 mg+SIM 125 mg (N=10) | SEL 18 mg+SIM 125 mg (N=10) | SIM 125 mg (N=10)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SEL 6 mg (N=20) | SEL 18 mg (N=22) | SEL 6 mg+SIM 125 mg (N=10) | SEL 18 mg+SIM 125 mg (N=10) | SIM 125 mg (N=10)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 0 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Infrequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 4 | 1 | 2 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Palatal swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 1 | 1
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 2 | 0 | 3 | 0
Hernia pain (General disorders) | 0 | 0 | 1 | 0 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site erythema (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2 | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 3 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 3 | 1 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2 | 1
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 1 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 1 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 7 | 1 | 2 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Euphoric mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 2 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years